CLINICAL TRIAL: NCT03089255
Title: Prospective Study to Assess the Foreseeable Impact of TIP Score on Thromboprophylaxis in Patients With Isolated Non-surgical Lower Limb Trauma Compared to the Physicians' Judgment in Standard Practice.
Brief Title: Assessment of the Impact of TIP Score on Thromboprophylaxis in Patients With Non-surgical Lower Leg Trauma.
Acronym: EvaTIP
Status: Completed | Type: Observational
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2017-A00291-52
Record Dates: First submitted 2017-03-17; First posted 2017-03-24 (Actual); Last update posted 2018-06-04 (Actual); Status verified 2018-06

CONDITIONS: Lower Limb Injury; Pulmonary Embolism; Venous Thromboses
Keywords: Thrombophylaxis; Deep Venous Thrombosis; Pulmonary Embolism; Lower Leg Trauma
MeSH Terms: conditions — Leg Injuries; Pulmonary Embolism; Venous Thrombosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Traumatic lesions are the leading causes of admission to the emergency center (39%), isolated non-surgical lower limbs trauma are in the foreground. Two recent meta-analyzes suggest the value of Low Molecular Weight Heparins (LMWH) which would reduce symptomatic Thromboembolism Events (TE) in patients with lower limb trauma. However, many recent studies conclude to the need of stratifying the TE risk according to the patient and the nature of his trauma to obtain an individualized therapeutic decision.

The retrospectively established L-TRIP (cast) score allows stratification of the risk without taking into account the type of trauma. The TIP score (Trauma, Immobilization and Patient) was established by consensus of international experts via the Delphi method.

We suggest that the application of the TIP score to rationalize indications of thromboprophylaxis in patients with isolated non-surgical trauma of a lower limb should reduce the rate of anticoagulation prescription without increasing the risk of symptomatic thromboembolic complications with a direct benefit for patients and medico-economic for the society.

DETAILED DESCRIPTION:
All patients admitted to the Emergency Departments for a nonsurgical isolated lower limb trauma necessitating rigid or semi-rigid immobilization, will be assessed for possible participation.

After the physicians had obtained the no-opposition of the patient, they will fill a questionnaire. This questionnaire includes the treatment chosen by the physician, the type of trauma, the type of immobilization chosen, and the patient's thromboembolic risk factors in order to calculate the TIP and L-TRIP (cast) scores retrospectively.

Phone follow-up will occur within 3 months to gather clinical event data (any signs of VTE, any bleeding events).

ELIGIBILITY:
Inclusion Criteria:

* Consultation in one of the emergency departments of the participating centres
* Isolated unilateral lower limb injury not requiring surgery
* Lower limb rigid or semi-rigid orthopedic immobilization (i.e. brace of plaster cast) for at least 5 days.
* Full insurance cover

Exclusion Criteria:

* Any anticoagulant or antiplatelet treatment prior to trauma
* Contra-indication to fondaparinux or LMWH
* Factors rendering 3-month follow-up impossible
* Imprisonment
* Inability to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients admitted in the Emergency Department for an isolated lower-leg trauma injury non surgical requiring semi-rigid or rigid immobilisation.
Sampling Method: Probability Sample
Enrollment: 196 (Actual)
Dates: Start 2017-04-03 (Actual); Primary Completion 2018-01-15 (Actual); Study Completion 2018-01-30 (Actual)

PRIMARY OUTCOMES:
Rate of prescriptions of prophylactic anticoagulation if TIP score was applied compared to the physicians' judgment in standard practice. | one day
  Compare two rate (percent) of prescription: obtained with standard practice and with the foreseeable TIP score calculated retrospectively.
  Score TIP is calculated retrospectively based on datas of the patients included. A threshold value is established by an expert consensus. A score is positive if it is higher than the threshold value, and negative if it is lower or equal to the threshold value. We consider that patients with a negative score would not have been treated by a prophylactic anticoagulation if the TIP score was applied.

SECONDARY OUTCOMES:
Rate of prescriptions of prophylactic anticoagulation if L-TRIP(cast) score was applied compared to the physicians' judgment in standard practice. | one day
  Compare two rate (percent) of prescription: obtained with standard practice and with the foreseeable L-TRIP(cast) score calculated retrospectively.
  A score is positive if it is higher than the threshold value, and negative if it is lower or equal to the threshold value. We consider that patients with a negative score would not have been treated by a prophylactic anticoagulation if the TIP score was applied.
The cumulative rate of symptomatic venous thromboembolism (i.e. deep venous thrombosis and/or pulmonary embolism) at 3 months from inclusion. | 3 months
  The following definitions are applied to confirm a suspected episode of symptomatic :
  * DVT: abnormal compression ultrasound
  * PE: an intraluminal filling defect in segmental or more proximal branches on spiral CT Scan or a perfusion defect of at least 75% of a segment with a local normal ventilation result (high-probability) on ventilation/perfusion lung scan or detected at autopsy.
The 3-month rate of major bleeding and of non-major clinically relevant bleeding according to the ISTH definition. | 3 months
  The safety endpoint is major bleeding, defined according to the recently published guidelines of the ISTH :
  1. Fatal bleed ing, and/or
  2. Symptomatic bleeding in a critical area or organ, such as intracranial, intraspinal, intraocular, retroperitoneal, intra- articular or pericardial, or intramuscular with compartment syndrome, and/or
  3. Bleeding causing a fall in hemoglobin level of 20 g.L (1.24 mmol.L) 1 or more, or leading to transfusion of two or more units of whole blood or red cells.
  The cumulative incidence of non-major clinically relevant bleeding. The cumulative incidence of minor bleeding.

CONTACTS AND LOCATIONS:
Overall Officials: Roy Pierre-Marie, MD, PhD, Principal Investigator — University Hospital, Angers
Locations (1):
- Douillet, Angers, France

IPD SHARING:
Plan to Share IPD: No